CLINICAL TRIAL: NCT01471054
Title: Dexamethasone Intravitreal Implant for Treatment of Macular Edema After Plaque Radiotherapy of Uveal Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not enroll enough patients.
Sponsor: Arman Mashayekhi (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Arman Mashayekhi, Principal Investigator, Assistant Professor, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wills IRB# 11-089
Record Dates: First submitted 2011-11-04; First posted 2011-11-11 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Macular Edema; Cystoid Macular Edema; Uveal Melanoma; Radiation Maculopathy; Radiation Retinopathy
Keywords: Plaque radiotherapy; Brachytherapy; Macular edema; Cystoid macular edema; Uveal melanoma; Radiation maculopathy; Radiation retinopathy; Ozurdex; Dexamethasone intravitreal implant
MeSH Terms: conditions — Macular Edema; Uveal Melanoma | interventions — Calcium Dobesilate; Dexamethasone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozurdex (Experimental): Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, measurement of best-corrected visual acuity (BCVA), complete eye examination, fundus photography, and optical coherence tomography. Fluorescein angiography will be repeated at 6 and 12 months. Each eye in the Ozurdex group can have a maximum total of three Ozurdex insertions at minimum of 4-month intervals in the first year after enrolling into the study.
  Interventions: Drug: Ozurdex
- Bevacizumab (Active Comparator): Patients will be followed at 1 week after the initial bevacizumab injection and then at 1,2, 3,4, 5, and 6 months after implant. Following the 6-month visit, the patients will be examined every 4-8 weeks depending on the status of their macular edema. At each visit patients will be checked for side effects of treatment, measurement of BCVA, complete eye examination, fundus photography, and optical coherence tomography. Fluorescein angiography will be repeated at 6 and 12 months. Eyes in the Bevacizumab group can have a maximum total of twelve (12) bevacizumab injections at minimum of 4-week intervals in the first year after enrolling into the study.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Ozurdex — Eyes in the Ozurdex group can have a maximum total of three Ozurdex insertions in the first 12 months after enrolling into the study. The criteria for retreatment with Ozurdex are:
  i.The study eye must have shown initial favorable response to prior Ozurdex implant (>10% decrease in central macular thickness with maintenance [change in BCVA of <=1 line] or improvement of visual acuity [increase of BCVA of >1 line]) ii. Interval since last Ozurdex implant should be > 4 and < 12 months. iii. The study eye must show definite evidence of recurrence of macular edema.
  Other Names: Dexamethasone intravitreal implant
  Arms: Ozurdex
Drug: Bevacizumab — Eyes in the Bevacizumab group can have a maximum total of twelve bevacizumab injections in the first year after enrolling into the study. All patients will receive 6 monthly injections after entering the study. After the sixth injection (at month 5) the interval between injections will be extended to 6 weeks if the study eye has shown initial favorable response to prior intravitreal bevacizumab.
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
To evaluate the safety and efficacy of dexamethasone intravitreal implant (Ozurdex) and compare it with safety and efficacy of intravitreal bevacizumab in eyes with macular edema after plaque radiotherapy of uveal melanoma.

DETAILED DESCRIPTION:
Plaque radiotherapy is a commonly used method for treatment of small and medium-sized uveal melanomas. Macular edema is one of the most common causes of visual loss after plaque radiotherapy and has been reported in up to 70% of patients with posterior uveal melanoma. Different methods have been proposed for treatment of post-radiation macular edema and include periocular steroid, intravitreal steroid, intravitreal vascular endothelial growth factor (VEGF) inhibitors, photodynamic therapy, and macular laser photocoagulation.

Injection of intravitreal triamcinolone (a form of steroid) has been found to be useful for treatment of different forms of macular edema but is associated with considerable rates of increased intraocular pressure (glaucoma). Dexamethasone is more potent than triamcinolone and can be safely injected directly into the vitreous cavity (intravitreal injection) but unfortunately its use in the form of intravitreal injection is not practical due to the short half-life of intraocular dexamethasone (about 3 hours).

Within the past several years, tiny drug delivery systems have been developed that allow sustained release of minute amounts of steroid into the back part (vitreous cavity) of the eye, when they are implanted into the vitreous cavity. Ozurdex is a biodegradable dexamethasone intravitreal implant that has been shown to be well-tolerated and effective for up to 6 months in reducing vision loss and improving visual outcome in eyes with different types of macular edema including those secondary to diabetic retinopathy and retinal vein occlusion.

In this study the investigators would like to evaluate the safety and effectiveness of Ozurdex (dexamethasone intravitreal implant) for treatment of macular edema developing after plaque radiotherapy of uveal melanoma.

ELIGIBILITY:
* Inclusion criteria:

  1. Patient age 18 years or more.
  2. Uveal melanoma treated with I-125 plaque radiotherapy.
  3. Visual acuity between 20/40 to 20/400 secondary to post-radiation macular edema.
  4. Central subfield retinal thickness > 300 micron.
  5. Duration of macular edema < 12 months.
  6. No potential contributing causes of decreased vision other than macular edema.
* Exclusion criteria:

  1. Visual acuity worse than 20/400 or better than 20/40.
  2. Monocular patient or poor vision in the non-study eye (<20/80).
  3. History of vitrectomy surgery.
  4. Panretinal photocoagulation or intraocular surgery within 3 months of enrollment.
  5. Concomitant or previous radiation optic neuropathy.
  6. Use of periocular, intravitreal, or systemic steroids within 6 month of enrollment in the study eye.
  7. Use of intravitreal VEGF antagonist within 6 weeks of enrollment.
  8. History of ocular hypertension or glaucoma, or intraocular pressure (IOP)>21 mmHg.
  9. History of steroid-induced glaucoma in either eye.
  10. Active ocular infection or history of herpetic eye infection.
  11. Clinically significant epiretinal membrane in the study eye.
  12. Iris neovascularization in the study eye.
  13. Clinically significant media opacity preventing acquisition of good-quality optical coherence tomography (OCT) in the study eye.
  14. Aphakia or anterior chamber intraocular lens.
  15. Poorly controlled diabetes (Hemoglobin A1c level >13%).
  16. Poorly controlled hypertension (Systolic pressure > 160 mm Hg or diastolic pressure > 90 mm Hg).
  17. Pregnancy (women of childbearing age should have negative pregnancy test and use contraception).
  18. Presence of any ocular condition that in the opinion of one of the investigators will prevent at least 2 lines of improvement in best-corrected visual acuity.
  19. Interval between plaque radiotherapy for uveal melanoma and intended date of dexamethasone intravitreal implant of less than 6 months.
  20. Evidence of activity or inadequate regression of the treated uveal melanoma after plaque radiotherapy (based on the judgment of the study investigators).
  21. Known allergy or hypersensitivity to any of the study medications or their components.
  22. History of prior myocardial infarction or stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Mashayekhi, MD, Principal Investigator — Wills Eye Hospital IRB Director
Locations (1):
- Ocular Oncology Service, Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shields CL, Cater J, Shields JA, Chao A, Krema H, Materin M, Brady LW. Combined plaque radiotherapy and transpupillary thermotherapy for choroidal melanoma: tumor control and treatment complications in 270 consecutive patients. Arch Ophthalmol. 2002 Jul;120(7):933-40. doi: 10.1001/archopht.120.7.933. PMID 12096964
- [Background] Horgan N, Shields CL, Mashayekhi A, Teixeira LF, Materin MA, Shields JA. Early macular morphological changes following plaque radiotherapy for uveal melanoma. Retina. 2008 Feb;28(2):263-73. doi: 10.1097/IAE.0b013e31814b1b75. PMID 18301032
- [Background] Horgan N, Shields CL, Mashayekhi A, Salazar PF, Materin MA, O'Regan M, Shields JA. Periocular triamcinolone for prevention of macular edema after plaque radiotherapy of uveal melanoma: a randomized controlled trial. Ophthalmology. 2009 Jul;116(7):1383-90. doi: 10.1016/j.ophtha.2009.01.051. Epub 2009 May 30. PMID 19481812
- [Background] Sutter FK, Gillies MC. Intravitreal triamcinolone for radiation-induced macular edema. Arch Ophthalmol. 2003 Oct;121(10):1491-3. doi: 10.1001/archopht.121.10.1491. No abstract available. PMID 14557194
- [Background] Gupta A, Muecke JS. Treatment of radiation maculopathy with intravitreal injection of bevacizumab (Avastin). Retina. 2008 Jul-Aug;28(7):964-8. doi: 10.1097/IAE.0b013e3181706302. PMID 18698298
- [Background] Bakri SJ, Beer PM. Photodynamic therapy for maculopathy due to radiation retinopathy. Eye (Lond). 2005 Jul;19(7):795-9. doi: 10.1038/sj.eye.6701637. PMID 15359269
- [Background] Hykin PG, Shields CL, Shields JA, Arevalo JF. The efficacy of focal laser therapy in radiation-induced macular edema. Ophthalmology. 1998 Aug;105(8):1425-9. doi: 10.1016/S0161-6420(98)98023-X. PMID 9709753
- [Background] Benhamou N, Massin P, Haouchine B, Audren F, Tadayoni R, Gaudric A. Intravitreal triamcinolone for refractory pseudophakic macular edema. Am J Ophthalmol. 2003 Feb;135(2):246-9. doi: 10.1016/s0002-9394(02)01938-4. PMID 12566041
- [Background] Martidis A, Duker JS, Greenberg PB, Rogers AH, Puliafito CA, Reichel E, Baumal C. Intravitreal triamcinolone for refractory diabetic macular edema. Ophthalmology. 2002 May;109(5):920-7. doi: 10.1016/s0161-6420(02)00975-2. PMID 11986098
- [Background] Scott IU, Flynn HW Jr, Rosenfeld PJ. Intravitreal triamcinolone acetonide for idiopathic cystoid macular edema. Am J Ophthalmol. 2003 Oct;136(4):737-9. doi: 10.1016/s0002-9394(03)00266-6. PMID 14516818
- [Background] Williams GA, Haller JA, Kuppermann BD, Blumenkranz MS, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Dexamethasone posterior-segment drug delivery system in the treatment of macular edema resulting from uveitis or Irvine-Gass syndrome. Am J Ophthalmol. 2009 Jun;147(6):1048-54, 1054.e1-2. doi: 10.1016/j.ajo.2008.12.033. Epub 2009 Mar 9. PMID 19268890
- [Background] Kuppermann BD, Blumenkranz MS, Haller JA, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled study of an intravitreous dexamethasone drug delivery system in patients with persistent macular edema. Arch Ophthalmol. 2007 Mar;125(3):309-17. doi: 10.1001/archopht.125.3.309. PMID 17353400
- [Background] Haller JA, Kuppermann BD, Blumenkranz MS, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled trial of an intravitreous dexamethasone drug delivery system in patients with diabetic macular edema. Arch Ophthalmol. 2010 Mar;128(3):289-96. doi: 10.1001/archophthalmol.2010.21. PMID 20212197
- [Background] Lowder C, Belfort R Jr, Lightman S, Foster CS, Robinson MR, Schiffman RM, Li XY, Cui H, Whitcup SM; Ozurdex HURON Study Group. Dexamethasone intravitreal implant for noninfectious intermediate or posterior uveitis. Arch Ophthalmol. 2011 May;129(5):545-53. doi: 10.1001/archophthalmol.2010.339. Epub 2011 Jan 10. PMID 21220619

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Afterwards, patients will be seen every 2 months. At each visit patients will undergo measurement of best-corrected visual acuity (BCVA), complete eye examination, fundus photography, and optical coherence tomography. Fluorescein angiography will be repeated at 6 and 12 months. Each eye in the Ozurdex group can have a maximum total of three Ozurdex insertions at minimum of 4-month intervals in the first year of study.
  The criteria for retreatment with Ozurdex are:
  i.The study eye must have shown initial favorable response to prior Ozurdex implant (>10% decrease in central macular thickness with maintenance [change in BCVA of <=1 line] or improvement of visual acuity [increase of BCVA of >1 line]) ii. Interval since last Ozurdex implant should be > 4 and < 12 months. iii. The study eye must show definite evidence of recurrence of macular edema.
- Bevacizumab: Patients will be followed at 1 week after the initial bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Afterwards, the patients will be examined every 4-8 weeks. At each visit patients will be checked for side effects of treatment, measurement of BCVA, complete eye examination, fundus photography, and optical coherence tomography. Fluorescein angiography will be repeated at 6 and 12 months. Eyes in the Bevacizumab group can have a maximum total of twelve (12) bevacizumab injections at minimum of 4-week intervals in the first year after enrolling into the study.
  All patients will receive 6 monthly injections after entering the study. After the sixth injection (at month 5) the interval between injections will be extended to 6 weeks if the study eye has shown initial favorable response to prior intravitreal bevacizumab.
Period: Overall Study
Arm/Group | Ozurdex | Bevacizumab
Started | 5 | 1
Completed | 1 | 1
Not Completed | 4 | 0
Not completed — Study terminated prematurely | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Afterwards, patients will be seen every 2 months. At each visit patients will undergo measurement of BCVA, complete eye examination, fundus photography, and optical coherence tomography. Fluorescein angiography will be repeated at 6 and 12 months. Each eye in the Ozurdex group can have a maximum total of three Ozurdex insertions at minimum of 4-month intervals in the first year of study.
  The criteria for retreatment with Ozurdex are:
  i.The study eye must have shown initial favorable response to prior Ozurdex implant (>10% decrease in central macular thickness with maintenance [change in BCVA of <=1 line] or improvement of visual acuity [increase of BCVA of >1 line]) ii. Interval since last Ozurdex implant should be > 4 and < 12 months. iii. The study eye must show definite evidence of recurrence of macular edema.
- Total: Total of all reporting groups
Arm/Group | Ozurdex | Bevacizumab | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66 [51 to 75] | 30 [30 to 30] | 60 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom Study Eye Showed >=2 Lines of Improvement in Best-corrected Visual Acuity
Description: The number of participants that developed 2 or more lines of visual acuity improvement in the study eye. Visual acuity was measured with Snellen eye chart placed 10 feet away from the patient.
Time Frame: At 12 months
Measure: Number; unit: participants
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 5 | 1
participants | 2 | 0

2. Secondary Outcome: Change in Central Subfield Retinal Thickness
Description: Increase or decrease in central subfield retinal thickness in microns based on spectral-domain optical coherence tomography measurement
Time Frame: At 12 months
Population: We were not able to measure central macular thickness at 12 months in one patient in the Ozurdex group due to advanced cataract.
Measure: Median (Standard Deviation); unit: micron
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for outcome of treatment, including change in central macular thickness.
- Bevacizumab: Patients will be followed at 1 week after intravitreal bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for outcome of treatment, including change in central macular thickness.
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 4 | 1
micron | -120 (231) | -4 (NA) — This group included only 1 patient and therefore standard deviation could not be calculated.

3. Secondary Outcome: Development of Glaucoma
Description: Intraocular pressure more than 21 mm Hg as measured with applanation tonometry.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including increased intraocular pressure.
- Bevacizumab: Patients will be followed at 1 week after intravitreal bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including increased intraocular pressure.
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 5 | 1
Participants | 3 | 0

4. Secondary Outcome: Development of Cataract
Description: Development of visually-significant lens opacity based on judgement of examining physician.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including cataract.
- Bevacizumab: Patients will be followed at 1 week after intravitreal bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including cataract.
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 5 | 1
Participants | 3 | 0

5. Secondary Outcome: Development of Retinal Detachment
Description: Development of rhegmatogenous retinal detachment in the study eye.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including retinal detachment.
- Bevacizumab: Patients will be followed at 1 week after intravitreal bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including retinal detachment.
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 5 | 1
Participants | 0 | 0

6. Secondary Outcome: Development of Vitreous Hemorrhage
Description: Development of hemorrhage in the vitreous cavity detectable with slit lamp examination or dilated funduscopy.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Ozurdex: Patients will be followed at 1 week after Ozurdex insertion (0.7 mg) and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including vitreous hemorrhage.
- Bevacizumab: Patients will be followed at 1 week after intravitreal bevacizumab injection and then at 1,2, 3,4, 5, and 6 months. Following the 6-month visit, patients will be seen every 2 months. At each visit patients will be checked for side effects of treatment, including vitreous hemorrhage.
Arm/Group | Ozurdex | Bevacizumab
Number analyzed (Participants) | 5 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ozurdex | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 0/5 | 0/1

LIMITATIONS AND CAVEATS:
Could not reach target number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No